CLINICAL TRIAL: NCT02864069
Title: Impact of Combined Behavioral Interventions on Cognitive Outcomes in MCI
Acronym: CBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Amy Jak, Associate Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NPSASA-14-321959
Record Dates: First submitted 2016-06-27; First posted 2016-08-11 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

ARMS (3):
- Walking Intervention (Experimental)
  Interventions: Behavioral: Walking Intervention
- Cognitive Training Intervention (Experimental)
  Interventions: Behavioral: Cognitive Training Intervention
- Combined Intervention (Experimental)
  Interventions: Behavioral: Combined Intervention

INTERVENTIONS:
Behavioral: Walking Intervention — The walking intervention will begin following baseline assessments and will be continued for 12 weeks. Participants will be given a pedometer to use daily and log their daily steps, with an identified goal of increasing step counts by 3000 steps a day over the course of the intervention. After obtaining a week long baseline step count, individuals in the intervention group will progressively increase their step counts by 100 steps daily each week for the first three weeks, by 200 steps daily for weeks four through six, by 300 steps daily for weeks seven through nine, and by 400 steps daily for weeks ten through twelve. Mean baseline step counts for sedentary older adults in our pilot work were 4150 per day; therefore, most participants will almost double their daily activity by the end of the intervention.
  Arms: Walking Intervention
Behavioral: Cognitive Training Intervention — In the CT condition, participants will use Brain HQ, a computer cognitive training program (Posit Science Corporation, San Francisco, CA), shown to be well tolerated by older adults with positive short- and long-term cognitive outcomes. Participants will use the program 60 minutes/day, 5 days/week for 12 weeks. If participants do not have a home computer/internet access, they can complete the modules at another location such as a public library, senior center, or at the MARC, but training will still be self-directed.
  Arms: Cognitive Training Intervention
Behavioral: Combined Intervention — The combined condition will concurrently follow both the walking and the CT programs as described above.
  Arms: Combined Intervention

SUMMARY:
Vast evidence supports use of physical exercise and cognitive stimulation for lowering risk for cognitive decline and dementia, with combinations of non-pharmacological interventions providing greatest promise for impacting cognitive aging. This, paired with limited cognitive benefits from pharmacological interventions in dementia, has shifted focus to non-pharmacological interventions administered earlier in the disease course. This application, therefore, proposes a randomized controlled trial (RCT; 12-week active intervention, 3- and 6-month follow-up) comparing 3 conditions: walking program (guided progressive increases in weekly step counts), computer-based cognitive training program (Brain HQ, Posit Science), and combination of the exercise and cognitive program, on cognitive, functional, and diagnostic outcomes in 60 sedentary, community-dwelling adults with mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* MCI diagnosis (can be self referral, will determine eligibility at baseline)

Exclusion Criteria:

* Dementia diagnosis
* Head trauma
* Neuro/psychiatric disorders
* Current substance dependence
* Sensory/mobility deficits
* No more than 1 hour of purposeful, aerobic activity/week
* Currently engaging in any other brain-stimulating computer program (No more than 1 hour a week)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Jak, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Walking Intervention | Cognitive Training Intervention | Combined Intervention
Started | 18 | 13 | 21
Completed | 12 | 5 | 13
Not Completed | 6 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking Intervention | Cognitive Training Intervention | Combined Intervention | Total
Number analyzed (Participants) | 18 | 13 | 21 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.06 (5.79) | 64.0 (4.06) | 69.48 (6.32) | 69.0 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 15 | 36
  Male | 7 | 3 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 12 | 20 | 50
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 18 | 8 | 20 | 46
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rivermead Behavioral Memory Test
Description: The Rivermead Behavioral Memory Test (RBMT) is an ecologically valid assessment of cognitive functioning that tests some skills specifically trained in the CT condition (e.g., name learning, and story learning) but also additional untrained skills such as prospective memory. Belongings subtest scaled scores: Minimum score = 1, Maximum score = 19; higher values represent better performance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Walking Intervention | Cognitive Training Intervention | Combined Intervention
Number analyzed (Participants) | 12 | 5 | 13
units on a scale | 11.08 (3.8) | 11.2 (2.95) | 12.31 (1.93)

2. Primary Outcome: Everyday Cognition Scale
Description: The Everyday Cognition Scale (ECog) assesses (via informant report) everyday cognitive functioning in memory, language, visuospatial, and executive functioning domains. Average total score was used: Minimum = 1, Maximum = 4, higher scores indicate greater impairment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Walking Intervention | Cognitive Training Intervention | Combined Intervention
Number analyzed (Participants) | 9 | 4 | 13
units on a scale | 1.50 (.64) | 1.14 (.17) | 1.24 (.30)

3. Primary Outcome: Older Peoples Quality of Life Questionnaire
Description: Self report assessment of quality of life specific to older adults. Assessment covers life overall, health, social relationships and participation, independence, control over life and freedom, home and neighborhood, psychological and emotional well-being, financial circumstances, leisure/activities, and culture and religion. Total score minimum = 35, max = 175; lower scores indicate better quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Walking Intervention | Cognitive Training Intervention | Combined Intervention
Number analyzed (Participants) | 12 | 5 | 13
units on a scale | 76.08 (20.74) | 72.20 (7.46) | 68.15 (16.01)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Walking Intervention | Cognitive Training Intervention | Combined Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/13 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/13 | 0/21
Other Adverse Events (participants affected / at risk) | 0/18 | 0/13 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT02864069/Prot_SAP_000.pdf